CLINICAL TRIAL: NCT06981611
Title: Vulvodynia Intervention (VI): the Effect of Multimodal Treatment for Provoked Vulvodynia
Brief Title: Vulvodynia Intervention: the Effect of Multimodal Treatment for Provoked Vulvodynia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karlstad University (Other)
Collaborators: Region Stockholm (Other Government); Region Örebro County (Other); Region Jönköping County (Other Government); Region Värmland (Unknown)
Responsible Party: Principal Investigator, Ida Flink, Professor in psychology, Karlstad University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-03946-01; 2023-00377 (Other Grant/Funding Number: Forte: Swedish Research Council for Health, Working Life and Welfare)
Record Dates: First submitted 2025-03-10; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Vulvodynia (Chronic Vulvar Pain)
Keywords: Vulvodynia; Provoked vulvodynia; multimodal treatment; cognitive behavioral therapy; cbt; couple treatment; single-case experimental design; sced; chronic pain; Vulvodynia Intervention
MeSH Terms: conditions — Vulvodynia; Color Vision Defects; Chronic Pain

STUDY DESIGN:
Intervention Model Description: The study utilizes a sequential single-case experimental AB design with randomized waiting period length (4, 5 or 6 weeks). Included in the design is also a pre-, post- and 6 month follow up measurement allowing for single group analysis of change. In addition, we collect qualitative data from patients, to explore experiences of participation in the study and the treatment.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to baseline length allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vulvodynia Intervention: a multimodal treatment for provoked vulvodynia (Experimental): A multimodal treatment consisting of approximately 11 treatment sessions, for provoked vulvodynia. Working with goal-directed behavior change that has both physiological and psychosocial components. The treatment sessions will be conducted with various professionals, via digital video meetings and meetings at the health care facilities. The first five sessions are conducted weekly, and the last six sessions are conducted biweekly. A follow-up session is conducted three months after the end of the treatment. Repeated measurements (twice a week) are being collected throughout this period.
  Interventions: Behavioral: Vulvodynia Intervention: a multimodal treatment for provoked vulvodynia
- Randomized to waiting period of 4, 5 or 6 weeks (No Intervention): Participants are randomized to a 4, 5 or 6 week waiting period/baseline. Repeated measurements (twice a week) are being collected throughout this period.

INTERVENTIONS:
Behavioral: Vulvodynia Intervention: a multimodal treatment for provoked vulvodynia — The intervention is based around physiological and psychosocial components working with goal-directed behavioral change. Includes both educational and practical elements, examples of these are vulva care, lubrication exercises, pelvic floor relaxation, work with thoughts, feelings, and behaviors related to the pain, as well as thoughts, feelings and behaviors related to sex and desire, and educational and practical elements focusing on open communication and validation. The treatment sessions are approximately 60 minutes each. There is a possibility for the participants to involve partner during two of the treatment sessions.
  Arms: Vulvodynia Intervention: a multimodal treatment for provoked vulvodynia

SUMMARY:
The purpose of this project is to develop and evaluate a multimodal treatment for provoked vulvodynia, by addressing the following specific research questions:

1. What is the feasibility and acceptability of this multimodal treatment protocol?
2. What are the effects on pain and psychosexual health?
3. How is the treatment perceived by patients, clinicians and stakeholders in the health care setting, and how do they view the possibilities for implementation?

Participants will be recruited through their health care unit and receive a multimodal treatment. The treatment consists of individual sessions with different professionals, in total 11 sessions over a time period of four months. It is possible to involve partners in the treatment during two of the treatment sessions. The majority of the sessions are digital video meetings but some are conducted at the health care unit. The treatment are based on physiological and psychosocial components that have previously shown positive effects for individuals with vulvodynia, and includes both educational and practical elements.

The participants will:

* Undergo a gynecological examination and a psychological assessment to determine if the treatment is suitable for their condition
* Undergo a multimodal treatment
* Complete questionnaires regarding their pain, physical tension, psychosexual and relational health and questions about the treatment
* Be asked to participate in an interview about their experience of the treatment and intimacy

DETAILED DESCRIPTION:
The study design consists of a mixed-methods design, where different methods are applied in the various sub-studies of the project.

Study 1, is an effectiveness evaluation, applying a sequential single case experimental AB design (SCED) with randomized baseline length, replicated across five healthcare contexts (n≈10-15 per unit, total N≈50-75).

Potential participants will be informed about the study at their health care unit and answer a few questions digitally to ensure that participation in the study is appropriate for them. An assessment will then be conducted and questions will be asked about the pain, psychological, sexual and relational health, and a diagnostic interview will be conducted to exclude other psychological issues that needs to be prioritized before vulvodynia treatment. After the assessment interview and inclusion, participants will be randomized to a 4, 5, or 6 week baseline period. Thereafter, the treatment will begin. During the baseline and treatment period, participants will complete a short self-assessment questionnaire, twice a week, to measure pain (primary outcome) and other key variables. To facilitate the repeated assessments, we will use the m-Path app, which was developed by KU Leuven University in Belgium to easily evaluate treatment for both patients and therapists. In addition to the repeated assessments, the treatment will be evaluated through a comprehensive web-based self-assessment questionnaire before and after the intervention and at a six-month follow-up, using the secure survey system called Survey and Report. through Karlstad university. The outcome measures are based on the ongoing work by the Swedish Agency for Health Technology Assessment and Assessment of Social Services.

Study 2, is a qualitative evaluation and initial assessment of the possibilities for implementing the treatment in the Swedish healthcare context.

Individual interviews with patients will be conducted and questions will be asked regarding their experience of the treatment model. Focus group interviews will be conducted with practitioners and questions will be asked regarding relevance, relative advantages, consistency with standard practices, usability, and adaptability. Since the treatment will be carried out in five healthcare units with different organizational and practical conditions, questions will specifically address unit-specific aspects that therapists and patients perceive as having facilitated or hindered the implementation and what could be improved in both treatment content and execution. The questions are based on the recommendations of the Swedish National Board of Health and Welfare and the Public Health Agency regarding the initial assessment of implementation possibilities.

To obtain the healthcare organization's perspective on implementation possibilities, interviews will be held with health care stakeholders within the participating healthcare units. These interviews will also focus on relevance, relative advantages, consistency with standard practices, usability, and adaptability.

The individual and focus group interviews will be conducted in person at the health care units or through digital video meetings. Data from focus group interviews and individual interviews will be recorded by audio, transcribed, and analyzed according to standard qualitative analysis methods, primarily inductive empirically driven Thematic Analysis (TA).

ELIGIBILITY:
Inclusion Criteria:

Biological sex: Female 18-40 years old Provoked vulvodynia

Exclusion Criteria:

* Severe psychological issues that should be prioritized before vulvodynia treatment (e.g., substance abuse, psychosis)
* Ongoing pregnancy
* Childbirth within the last year
* Post-traumatic stress disorder (PTSD) related to sexual trauma
* Insufficient mastery of the Swedish language
* No experience of vaginal sex, as vaginismus might be suspected, which requires different treatment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain during touch and/or insertion of an object | Pre, post treatment (25 weeks after the baseline measurement started) and at 6 month follow-up, during baseline (4, 5 or 6 weeks) and treatment period measured twice a week for 25 weeks.
  Provoked pain during sexual and non-sexual activities. Seven activities where pain is rated on a scale from 0 to 10. Higher scoring indicates higher degree of pain. There are also subsequent questions regarding whether they have performed the described activity or not within a specific time frame.

SECONDARY OUTCOMES:
Change in sexual function | Pre and post treatment (25 weeks after the baseline measurement started) and at 6 months follow-up
  The Female Sexual Function Index (FSFI) is a self-report measure of female sexual function that assesses six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. It consists of 19 questions, rated on a 5-point scale, with a higher score indicating a better sexual function.
Change in treatment goal attainment | Pre, post treatment (25 weeks after the baseline measurement started) and at 6 month follow-up. Repeated measures twice a week during baseline (4, 5 or 6 weeks) and treatment period, for 25 weeks.
  Participants chose an individual treatment goal and rate treatment goal attainment, from 0-10, 0= the goal is not at all achieved, 10= the goal is achieved.
Change in pelvic floor tension | Pre, post treatment (25 weeks after the baseline measurement started) and at a 6 month follow-up. During baseline and treatment period measured twice a week, for 25 weeks.
  Self-report assessment of pelvic floor tension and pelvic floor relaxation. Two items rated on a 11-point scale, from 0-10, higher scores indicate greater tension and more difficulty relaxing the pelvic floor, and physiotherapeutic examination.
Change in sexual satisfaction | Pre and post treatment (25 weeks after the baseline measurement started) and at 6 months follow-up
  Global measure of sexual satisfaction (GMSEX), 5 items rated on a 7-point scale. Higher scores indicate a higher degree of sexual satisfaction.
Change in interpersonal and self focused sexual goals | Pre and post treatment (25 weeks after the baseline measurement started), and at 6 months follow-up
  Approach avoidance sexual goals (AASQ), self focused sexual goals and interpersonal sexual goals, 23 items rated on a 7-point scale, participants rates the importance of self focused or interpersonal reasons, influencing why they typically engage in sex. Higher scores indicates greater importance.
Change in perceived intimacy | Pre and post treatment (25 weeks after the baseline measurement started), and at 6 months follow-up
  9 items regarding self and partner disclosure, partner responsiveness and closeness, rated on a 7-point scale, with higher scores indicating greater perceived intimacy.
Change in life interference, sexual function interference and impact on relationship | Pre and post treatment (25 weeks after the baseline measurement started) and at 6 months follow-up
  Vulvar pain assessment questionnaire (VPAQ) Inventory is a disease-specific set of measurement scales to capture the biopsychosocial nature of vulvodynia. We are using the parts from the questionnaire that evaluates life interference, sexual function interference, impact on relationship and sexual communication.
  Life interference: 11 items rated on a 6-point scale from 0 (not at all) to 4 (avoid because of pain). Higher scores indicating greater life interference.
  Sexual function interference: 10 items rated on a 6-point scale from 0 (not at all) to 4 (avoid because of pain)
  Impact on relationship: 6 items about intimacy and, general and sexual communication rated on a 5-point scale from much worse to much better. Higher scoring indicates that the vulva pain has lower impact on the relationship.
  6 items about communication with partner rated on a 5-point scale from 0 (largely uncomfortable) to 4 (largely comfortable). Higher scoring indicates
Change in depressive symptoms | Pre and post treatment (25 weeks after the baseline measurement started) and at 6 months follow-up
  Using the patient health questionnaire (PHQ-9), 9 items are rated on a 4-point scale, from 0 to 3. Higher scores indicating higher degree of depression symtoms.
Change in anxiety symptoms | Pre and post treatment (25 weeks after the baseline measurement started) and at 6 months follow-up
  Using the Generalized Anxiety Disorder questionnaire (GAD-7), 7 items rated on a 4-point scale from 0 to 3, higher scoring indicating a higher degree of anxiety symptoms.
Change in quality of life | Pre and post treatment (25 weeks after the baseline measurement started) and at 6 months follow-up
  World Health Organization Quality of Life-BREF, 1 item where participants rates their quality of life, on a 5-point scale from 1 to 5, higher scoring indicating greater quality of life.

OTHER OUTCOMES:
Evaluation of how much time participants spend on the treatment and related exercises | during treatment period
Demographic | Pre treatment (25 weeks after the baseline measurement started). Questions about partner/-s are measured pre and post treatment (25 weeks after the baseline measurement started) and at 6 month follow-up.
  Age, country of birth, educational level, occupation, if they have a partner/-s, how long they have been in that relationship/-s, gender of partner/-s, if they have kids, childbirth during the last year, ongoing pregnancy, menstruation
Change in sexual desire and arousal | Repeated measure twice a week during baseline and treatment period, for 25 weeks.
  Two items from the female sexual function index, measuring sexual desire and arousal, rated on a 5-point scale. Higher scoring indicate greater sexual desire and arousal.
Change in pain catastrophizing | Pre and post treatment (25 weeks after the baseline measurement started) and at 6 months follow-up
  Pain catastrophizing scale (PCS) evaluates participants negative cognitive and emotional reactions to pain. It assesses the extent of catastrophic thinking due to pain according to three subscales: rumination, magnification and helplessness. 13 items rated on a 5-point scale from 0 (not at all) to 4 (all the time). Higher scores indicating greater levels of pain catastrophizing.
Change in avoidance and endurance related to sexual activities | Repeated measure twice a week during baseline and treatment period, for 25 weeks
  Two items from the CHAMP Sexual Pain Coping Scale (CSPCS), rated on a 7-point scale, with higher scores indicating a higher degree of avoidance and endurance.
Experiences of sexual and physical abuse | Pre treatment
  Using the Sexual and Physical Abuse Questionnaire (SPAQ). 8 questions about experiences of sexual and physical abuse.
Treatment expectations | Pre treatment
  2 items rated on a 11-point scale, from 0 to 10. Higher scoring indicating higher expectations that this treatment will be helpful.
Negative treatment effects | Post treatment (25 weeks after the baseline measurement started)
  1-2 items measuring negative effects of the treatment. One questions that asks if the participant experienced any negative effects of the treatment, with a following question asking the participant to describe more in an open answer.
Perceived treatment improvement and satisfaction | Post treatment (25 weeks after the baseline measurement started)
  4 items rating potential improvement and satisfaction on a 6-point scale (1-6), higher scoring indicating greater improvement and satisfaction.
Change in sexual pain coping | Pre and post treatment (25 weeks after the baseline measurement started) and at 6 months follow-up
  Using items from the CHAMP Sexual Pain Coping Scale, 12 items assess coping strategies for sexual pain: avoidance and endurance, rated on a 7 point-scale from 1 to 7, where higher scoring indicating a higher degree of avoidance and/or endurance.
Experience of treatment | Post treatment (25 weeks after the baseline measurement started)
  Semi structured interviews, individual interviews and focus groups, probing qualitative aspects of the treatment experience, and the experience of implementation of patients, treating practitioners and clinical managers.

CONTACTS AND LOCATIONS:
Locations (1):
- Karlstad University, Karlstad, Sweden

IPD SHARING:
Plan to Share IPD: No
Because of the sensitive nature of the data. Data can be provided by request.